CLINICAL TRIAL: NCT00319241
Title: Relational Parenting Group for Opioid-addicted Mothers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: APT Foundation, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Nancy E Suchman, PhD, Yale University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9401007365; R01DA011498 (NIH)
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2008-06

CONDITIONS: Substance Abuse; Child Abuse
Keywords: parenting intervention; substance abuse treatment; mother-child relations; parent-child relations; child abuse and neglect
MeSH Terms: conditions — Substance-Related Disorders

INTERVENTIONS:
Behavioral: Parenting Intervention

SUMMARY:
This study is a randomized trial of interventions to improve parent-child relationships of drug-dependent mothers.

DETAILED DESCRIPTION:
In this Stage II study, we will conduct a randomized clinical trial of the Relational Parenting Mothers' Group (RPMG), an intervention designed for opioid abusing mothers with children between the ages of 7 and 14 which was manualized and tested as part of a Stage I study (NIDA # P50-DA09241; September 1, 1994- August 31, 1997). This intervention was developed in recognition of the substantial psychosocial risks faced by substance abusing mothers and their offspring, and the notable lack of parenting interventions currently available for addicted mothers with children past the preschool years. Based on developmental psychopathology perspectives on resilience, this integrative treatment addresses multiple levels of adversity (individual, family, and community) faced by addicted mothers: risks that typically result in negative parenting behaviors and psychosocial distress among the mothers and concomitantly, psychiatric disturbance among their offspring. Designed as a supplement to standard drug counseling, RPMG is a structured and time-limited treatment, entailing 24 weekly group sessions of 1½ hours each.

Preliminary data collected in the Stage I pilot study have attested to the promise of RPMG in terms of diverse parenting behaviors and psychiatric outcomes among both mothers and their children. In the proposed study, we will conduct a randomized clinical trial in which mothers receiving RPMG as a supplement to Recovery Training (RT, a manualized group intervention representing standard drug counseling offered in methadone clinics) will be compared with those who receive RT alone. The RPMG clinical team will include one masters/doctoral level therapist and one assistant therapist and RT groups will be conducted by drug counselors; all therapists (RPMG & RT) will be trained and supervised by our research team. One hundred sixty mothers will be randomized to one of the two treatment conditions. Multiple-method, multiple-informant assessments will be used to measure salient outcomes; these will include reports from mothers and their children, and from the mothers' clinicians and their children's teachers.

We will address the following specific aims in this study:

1. We will evaluate the effectiveness of the Relational Parenting Mother's Group (RPMG) as a supplement to Recovery Training (RT) vs. Recovery Training alone in terms of a) mothers' parenting behaviors, b) their psychosocial adjustment, c) their children's psychosocial adjustment, and d) mothers' treatment compliance.
2. We will evaluate the comparative durability of RPMG+RT vs. RT in terms of the outcomes in Aim #1, and in terms of delayed improvement in frequency of illicit drug use, HIV-risk behaviors, and other problems related to drug use.
3. We will examine how specific maternal characteristics interact with treatment to affect outcomes. Guided by previous research, these characteristics will include mothers' intelligence, readiness for change, and sensation seeking.

ELIGIBILITY:
Inclusion criteria:

* female adult humans
* enrollment in methadone treatment for opioid addiction
* caring for a child between the ages of 7 and 14 years

Exclusion Criteria:

* suicidality/homicidality requiring more intensive level of care
* serious cognitive impairment (AIDS-related dementia or schizophrenia)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 1998-01; Primary Completion 2003-10 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Mother's risk for maltreating her child
Mother's affective and instrumental parenting
Mother's psychosocial adjustment

SECONDARY OUTCOMES:
Children's psychosocial adjustment
Mother's substance abuse

CONTACTS AND LOCATIONS:
Overall Officials: Suniya Luthar, Ph.D., Principal Investigator — Teachers College, Columbia University; Nancy Suchman, Ph.D., Study Director — Yale University
Locations (1):
- The APT Foundation, New Haven, Connecticut, United States

REFERENCES:
- [Result] Luthar SS, Suchman NE, Altomare M. Relational Psychotherapy Mothers' Group: a randomized clinical trial for substance abusing mothers. Dev Psychopathol. 2007 Winter;19(1):243-61. doi: 10.1017/S0954579407070137. PMID 17241493